CLINICAL TRIAL: NCT06778850
Title: A Randomized, Double-blind, Placebo-controlled Phase I/IIa Clinical Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Ascending Doses of MDR-001 Tablets Administrated Orally in Healthy Participants and Obese/ Overweight Participants
Brief Title: A Phase I/IIa Clinical Study to Assess the Single and Multiple Ascending Doses of MDR-001 Tablets in Healthy Participants and Obese/ Overweight Participants
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MindRank AI Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MDR-001-CN-01
Record Dates: First submitted 2025-01-07; First posted 2025-01-16 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-01

CONDITIONS: Overweight and Obese Volunteers
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MDR-001（SAD） (Experimental): Single doses of MDR-001 administered orally.
  Interventions: Drug: MDR-001
- Placebo (SAD) (Experimental): Placebo administered orally.
  Interventions: Drug: palcebo
- MDR-001 (MAD) (Experimental): Multiple doses of MDR-001 administered orally.
  Interventions: Drug: MDR-001
- Placebo (MAD) (Experimental): Placebo administered orally.
  Interventions: Drug: palcebo

INTERVENTIONS:
Drug: MDR-001 — Oral administration of small molecule MDR-001 tablets
  Arms: MDR-001 (MAD); MDR-001（SAD）
Drug: palcebo — Administered orally placebo
  Arms: Placebo (MAD); Placebo (SAD)

SUMMARY:
To investigate the safety and tolerability after single and multiple ascending doses of MDR-001 Tablets administered orally in healthy participants and obese/ overweight participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are aged ≥ 18 and ≤ 55 years at the time of signing the informed consent; no gender restriction.
* Participants with 27 ≤ body mass index (BMI) ≤ 45 kg/m2.
* For male participants, a waist circumference ≥ 90 cm is required, while female participants ≥ 85 cm.

Exclusion Criteria:

* Participants with any condition that increases the risk of bleeding, such as hemorrhoids, acute gastritis, or gastric and duodenal ulcers.
* Participants with personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia 2 (MEN2), or those with hereditary diseases that easily induce to medullary thyroid carcinoma.
* Participants with a history of pancreatitis or symptomatic gallbladder disease.
* Serum calcitonin > ULN at screening.
* Participants with systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg at screening.
* Participants with ALT >2 × ULN and /or AST > 2 × ULN at screening.
* Participants whose fasting triglycerides > 5.7 mmol/L, total cholesterol > 7.75 mmol/L, low-density lipoprotein cholesterol > 4.9 mmol/L at screening.
* Participants with abnormal uric acid levels accompanied by clinical symptoms (those without clinical symptoms can be included).
* Participants with fasting blood glucose levels > 7 mmol/L.
* Participants with creatinine clearance < 60 mL/min at screening [calculation formula: CLcr: (140 - age) × weight (kg) / [72 × 0.0113 × Scr (μmol/L)], × 0.85 for females].
* Participants have experienced significant changes in diet or exercise habits or within ≥5% changes in body weight within 3 months prior to screening.
* Participants with clinically significant ECG abnormality deemed unsuitable participation for study by the investigator; or with ECG QTcF values > 450 ms for male participants or > 470 ms for female participants.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 131 (Estimated)
Dates: Start 2023-06-09 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through Day 84
  A summary of TEAEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
PK: Area Under the Concentration Versus Time Curve (AUC) of MDR-001 | Baseline through Day 84
  PK: AUC of MDR-001
Change from Baseline in Fasting Glucose | Baseline through Day 84
  Change from Baseline in Fasting Glucose
Pharmacokinetics (PK): Maximum Concentration (Cmax) of MDR-001 | Baseline through Day 84
  PK: Cmax of MDR-001
Change from Baseline in Glycated Hemoglobin (HbA1c) | Baseline through Day 84
  Change from Baseline in HbA1c
Change from Baseline in Body Weight | Baseline through Day 84
  Change from Baseline in Body Weight

CONTACTS AND LOCATIONS:
Locations (1):
- The first hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No